CLINICAL TRIAL: NCT05759312
Title: Zimberelimab Combined With Metformin in the Treatment of Recurrent Ovarian Clear Cell Carcinoma: A Pilot Study
Brief Title: Zimberelimab Plus Metformin for Recurrent Ovarian Clear Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Libing Xiang, Associate chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zsfud-OC-001
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Clear Cell Carcinoma
Keywords: Ovarian Clear Cell Carcinoma; Immune Checkpoint Inhibitor; Metformin
MeSH Terms: interventions — zimberelimab; spartalizumab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zimberelimab plus metformin (Experimental): Patients will start metformin at 1,000mg by mouth once daily during a 7-day induction period prior to starting zimberelimab. The dose will be increased by 500mg every 7 days until reaching the target dose of 2000mg. Zimberelimab will be administered at a fixed dose of 240 mg IV every 14 days. Treatment will continue until disease progression confirmed by RECIST criteria v1.1, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Zimberelimab; Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Zimberelimab — Zimberelimab 240mg IV every 2 weeks
  Other Names: Anti PD-1
Drug: Metformin Hydrochloride — Metformin 2000mg PO QD
  Other Names: Metformin

SUMMARY:
This study aims to evaluate the safety and effectiveness of zimberelimab combined with metformin in treating relapsed/persistent ovarian clear cell carcinoma.

DETAILED DESCRIPTION:
Ovarian clear cell carcinoma (OCCC) is one of the rare subtypes of ovarian cancer, yet its prognosis is extremely poor. Previous studies indicate that PD-1 inhibitors may have clinical benefits for OCCC patients. This single-arm, single-center, pilot study evaluates the safety and effectiveness of zimberelimab combined with metformin in treating relapsed/persistent ovarian clear cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years to ≤ 75 years
* Pathologic confirmed ovarian clear cell carcinoma
* Patients with recurrent or persistent ovarian clear cell carcinoma must have at least one-line pretreated platinum-containing chemotherapy
* According to the definition of RECIST1.1, the patient must have measurable lesions
* PD-L1 Combined Positive Score ≥ 1
* ECOG performance status of 0 to 2
* Adequate bone marrow, liver, and renal function to receive combined immunotherapy
* Written informed consent

Exclusion Criteria:

* Histological evidence of non-ovarian clear cell carcinoma
* Lack of tumor samples (archived and/or recently obtained)
* Previous administration of immunotherapy
* Patients have been vaccinated with the live vaccine or received anti-tumor treatment within 4 weeks before the first administration
* An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) within 2 years before the first administration
* Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ or breast cancer (without any signs of relapse or activity) Symptomatic or uncontrolled visceral metastases that require simultaneous treatment
* Patients are known to be allergic to the active ingredients or excipients of zimberelimab or metformin
* Known human immunodeficiency virus (HIV) infection history (HIV 1/2 antibody positive).
* Untreated active hepatitis B (defined as HBsAg positive and the number of copies of HBV-DNA detected at the same time is greater than the upper limit of the normal value of the laboratory department of the research center)
* Contraindications to metformin: kidney dysfunction or abnormal creatinine from any cause; acute or metabolic acidosis

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  The proportion of patients with complete response (CR) and partial response (PR) assessed by the investigator in accordance with the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years
  The time from entry into the study to the diagnosis of the first progression or recurrence or death, whichever occurs first
Overall survival | Up to 2 years
  The time from date of randomization until the date of death from any cause or last follow-up
Disease control rate | Up to 2 years
  The proportion of patients who achieved complete response (CR) or partial response (PR) or stable disease (SD) assessed by the investigator in accordance with the RECIST 1.1 criteria
Duration of response | Up to 2 years
  The time interval from the first record of disease response to disease progression or death (whichever occurs first)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 2 years
  The adverse event assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Patterns of subsequent recurrence | Up to 2 years
  The number and sites of subsequent recurrence, including pelvic, abdominal, retroperitoneal lymph nodes, hepato-celiac lymph nodes and distant metastases and ascites, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Libing Xiang, Principal Investigator — Department of Gynecologic Oncology, Zhongshan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: No